CLINICAL TRIAL: NCT03213418
Title: Electroretinogram: a New Human Biomarker for Smoking Cessation Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to delay in recruitment during COVID and cost considerations, the study will need to end without meeting its recruitment target and meeting compliance requirements.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Sean Luo, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 7519
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Smoking Cessation; Tobacco Use; Tobacco Dependence; Tobacco Use Disorder; Tobacco Smoking; Cigarette Smoking; Nicotine Dependence; Nicotine Use Disorder; Smoking; Smoking, Cigarette
Keywords: tobacco; smoking; Tobacco Use; Tobacco Dependence; Smoking, Tobacco; Cigarette Smoking; Cigarette; Nicotine
MeSH Terms: conditions — Smoking Cessation; Tobacco Use; Tobacco Use Disorder; Tobacco Smoking; Cigarette Smoking; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contingency management (Experimental)
  Interventions: Behavioral: Contingency management

INTERVENTIONS:
Behavioral: Contingency management — Contingency management is an evidence-based psychotherapy program that promotes behavioral change with financial incentives.

SUMMARY:
This project aims to develop electroretinogram as a new putative marker for dopamine release, and as a predictor of treatment response among patients seeking treatment for smoking cessation. Tobacco smoking continues to be a major public health challenge. Dopamine is a neurotransmitter released in the brain. Several lines of evidence suggest that dopamine release deficit in the brain is involved in the development and maintenance of nicotine dependence. The investigators hypothesize that smokers who do not have a deficit in dopamine release will more readily respond to behavioral treatment for smoking cessation, and in particular, financial incentives contingent on abstinence (Contingency Management). Previous pilot data suggest electroretinogram (ERG), which records electrical signals from the retina in response to light, is a clinically accessible correlate to dopamine release in the brain. The project proposes an ERG-based biomarker, and a pilot clinical trial to apply this biomarker to personalize smoking cessation treatment. This clinically tractable biomarker of central dopamine release may have a large number of future applications in the diagnosis and treatment of other mental illnesses and substance use disorders.

The study will recruit normal controls and smokers, measure ERG before and after a standard dose of oral immediate release methylphenidate. Smokers will undergo a 12-week standardized treatment course of CM. The investigators will test whether smoking status and the response to CM are correlated to changes in ERG in response to methylphenidate challenge.

ELIGIBILITY:
Inclusion Criteria

1. Be between the ages of 18 to 55 years of age.
2. Have an estimated average daily consumption of greater than 10 cigarettes.
3. Have a Fagerstrom Nicotine Dependence Scale (FTND) >= 5.
4. Is willing to try a method of smoking cessation without using any pharmacologic help for 3 months.

Exclusion Criteria

1. Present with a serious psychiatric illness or substantial suicide or violence risk, as assessed by a licensed clinician involved in the screening phase of the study.
2. Present with any history or current substance use disorder (other than tobacco use disorder), or significant substance use for any substance other than nicotine, alcohol or caffeine, defined as greater than once weekly use.
3. Legally mandated to complete a substance abuse treatment program.
4. Express a desire or intent to obtain additional substance abuse treatment while in the study.
5. Have history of psychotic symptoms such as hallucinations and delusions.
6. Have history of using other smoking cessation treatment, either psychotherapeutic or pharmacologic, in the past 2 months.
7. Have history of any chronic medical or ophthalmologic diseases that may affect retinal function (including but not limited to diabetes, age related macular degeneration, retinitis pigmentosa, narrow angle glaucoma, or neurological conditions, such as Parkinson's disease) and that may affect ERG recordings.
8. The use of any prescription or over the counter medication that may affect the retinal dopamine system, including bromocriptine, antipsychotics, or anticholinergics.
9. If female, be currently pregnant, breastfeeding, or lack of effective birth control during 15 days prior to before the ERG.
10. The use of stimulant medications in the past 12 months.
11. Have a known hypersensitivity to stimulant medications
12. Have history of medical condition that contraindicates the use of methylphenidate, including any history of significant cardiovascular disease or abnormal screening EKG.
13. Is unable to understand or consent to study procedure, or is in the opinion of the study clinician to be unlikely to be able to tolerate the study treatment procedure.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Abstinence | 1 month
  Prolonged abstinence from cigarette smoking will be measured through a combination of self-reported timeline follow back, as it is corroborated with urine cotinine and expired CO levels.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Luo, MD, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- NYSPI, STARS Clinic, 3 Columbus Circle, suite 1408, 14th Floor, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will determine feasibility of IPD depending on resource allocation.